CLINICAL TRIAL: NCT01357408
Title: Phase 4 Registry Study Will Evaluate the Ability of Cardiac Rhythm (Cardiac Compass) Data to Predict Future Cardiac Events in Heart Failure (HF) Patients Recently Discharged After a Hospitalization for Heart Failure Who Have or Plan to Have a Implanted Loop Recorder (ILR), Specifically, the Reveal XT Device.
Brief Title: Heart Failure and Risk of Re-Admissions Determined by Abnormal REVEAL Parameters
Acronym: HF-RADAR
Status: Terminated | Type: Observational
Why Stopped: enrollment futility
Sponsor: Thomas Jefferson University (Other)
Collaborators: Central Bucks Specialists, Ltd. (Other); Drexel University (Other); The Valley Hospital (Unknown); Saint Thomas Research Institute, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 080-18014-J66601
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Heart Failure
Keywords: without an indication for ICD or CRT; left ventricular function greater than or equal to 40%
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- REVEAL XT device: Subjects implanted at time of admission for HF or to be implanted within 14 days of discharge from HF hospitalization for clinical indications>

SUMMARY:
The purpose of the Heart Failure and Risk of re-Admissions Determined by Abnormal REVEAL Parameters (HF RADAR) study is to evaluate the ability of cardiac rhythm (Cardiac Compass) data to predict future cardiac events in heart failure (HF) patients recently discharged after a hospitalization for heart failure who have or plan to have a implanted loop recorder (ILR), specifically, the Reveal XT device. The study will enroll 40 HF patients (with LV function ≥ 40%) admitted to an acute care facility (observation status or hospital stay) for heart failure who either have a Reveal XT device in place or plan to have the ILR device inserted for clinical indication within 14 days of discharge from the hospitalization. HF patients will be followed for 6 months. Device date will be captured during normal clinic visits and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant/non lactating women ≥ 18 years.
2. Admission to hospital or observation unit for worsening heart failure.
3. Has a Reveal XT device or has plans for a device implant for a clinical indication within 14 days of discharge.
4. Ejection fraction ≥40% by echocardiogram within 6 months of enrollment
5. Able to participate in the study for at least 6 months.
6. Not currently enrolled in another study.
7. Able to provide informed consent and complete scheduled study visits.

Exclusion Criteria:

1. Has a clinical indication for a therapeutic cardiac device (pacemaker or defibrillator)
2. History of permanent atrial fibrillation or atrial flutter.
3. History of uncontrolled hypertension (high blood pressure)
4. Has a previously implanted cardiac device (pacemaker or defibrillator) in place.
5. Stage IV or V chronic renal dysfunction (estimated GFR <25 ml/min per 1.73 m2)
6. End-stage (Stage D) HF, including chronic ionotropic drugs infusions or left ventricular assist device
7. Waiting on the transplant list as an UNOS status 1A or 1B patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HF patients (with LV function ≥ 40%) admitted to an acute care facility (observation status or hospital stay) for heart failure who either have a Reveal XT device in place or plan to have the ILR device inserted for clinical indication within 14 days of discharge from the hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Worsening HF symptoms or HF-related clinical events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States